CLINICAL TRIAL: NCT05961735
Title: Comparison of PECS II Block and Combined Serratus Anterior Plane Block to Reduce Acute Pain After Mastectomy
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf Özgüner, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: AnkaraEtlikYusufOzguner004
Record Dates: First submitted 2023-07-14; First posted 2023-07-27 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative
Keywords: PECS II Block; Combined Serratus Anterior Plane Block; Mastectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with PECS II Block: PECS 2 block will be applied to patients in this group.
  Interventions: Other: PECS II Block
- Patients with Combined Serratus Anterior Plane Block: Combined Serratus Anterior Plane Block will be applied to patients in this group.
  Interventions: Other: Combined Serratus Anterior Plane Block

INTERVENTIONS:
Other: PECS II Block — The Pecs II block is applied to the patients after induction of anesthesia .
  Groups: Patients with PECS II Block
Other: Combined Serratus Anterior Plane Block — Combined Serratus Anterior Plane Block is applied to the patients after induction of anesthesia .
  Groups: Patients with Combined Serratus Anterior Plane Block

SUMMARY:
In this study, PECS II block or CSAB will be applied to patients who have had a modified radical mastectomy under general anesthesia for postoperative pain relief by using 30 ml of 0.25% bupivacaine .All patients will receive tramadol with a patient-controlled analgesia device during the postoperative period. Pain, nausea-vomiting, additional analgesic and antiemetic drug requirement, within 24 hours postoperatively will be compared between groups.

In this study, it was aimed to compare the efficacy of both peripheral nerve block methods in patients after mastectomy.

DETAILED DESCRIPTION:
Breast cancer ranks first among the most common malignant neoplasms in women. Surgery has been a mainstay of breast cancer treatment for several decades and historically, a modified radical mastectomy was the primary method of treatment for breast cancer. Poorly controlled acute postoperative pain is associated with increased morbidity, functional and quality-of-life impairment. Additionally, severe acute postoperative pain is found to be a risk factor for chronic pain.

Thoracic paravertebral, thoracic epidural, intercostal nerve, and interscalene brachial plexus blocks have been used for anesthesia and abirritation during modified radical mastectomy, but their application is limited due to the complex nature of the procedures and serious complications. There is growing interest in the pectoralis nerve (PECS) blocks and serratus anterior block (SAB) which are less invasive as an analgesic technique during breast surgeries to reduce postoperative pain.

The Pecs I block is a single injection of local anaesthetic between pectoralis major and pectoralis minor muscles at the level of the 3rd rib to anaesthetise the lateral and medial pectoral nerves. The Pecs II block is a modified Pecs I block and can be achieved with one needle insertion point. Local anaesthetic is placed between pectorals major and minor as for a Pecs I block and then between pectoralis minor and serratus anterior muscles.

Numerous clinical studies focusing on the analgesic potential of PECS block in breast augmentation surgery, small breast surgery and breast cancer surgery have yielded positive results. SAD is more superficial, easy to access and less likely to have complications like PECS block. SAPB can be implemented in two ways. Deep SAB (DSAB) is applied under the serratus anterior muscle, while superficial SAB (YSAB) is applied over the serratus anterior muscle. In recent years, deep and superficial SAB, that is, combined SAB (CSAB), has been started to be applied in order to increase the effect area of local anesthetics and to prevent block failure.

In this study, PECS II block or CSAB will be applied to patients who have had a modified radical mastectomy under general anesthesia for postoperative pain relief by using 30 ml of 0.25% bupivacaine .All patients will receive tramadol with a patient-controlled analgesia device during the postoperative period. Pain, nausea-vomiting, additional analgesic and antiemetic drug requirement, within 24 hours postoperatively will be compared between groups.

In this study, it was aimed to compare the efficacy of both peripheral nerve block methods in patients after mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-80
* Patients with ASA score I-II-III
* Patients with a body mass index (BMI) between 18 and 40
* Patients who underwent PECS-II block or CSAB with mastectomy in the operating room

Exclusion Criteria:

* Patients under the age of 18 and over the age of 80
* Patients with an ASA score of IV and above
* Patients with advanced co-morbidity
* Patients with a history of bleeding diathesis
* Patients who have infection in the area which is to be blocked
* BMI below 18 and over 40
* Patients undergoing emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who undergone mastectomy surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Pain on the Numeric Rating Scale (NRS) | 0 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 2 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 4 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 8 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 12 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 24 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.
Total opioid consumption | 24 hours postoperatively
  All patients will receive tramadol with a patient-controlled analgesia device during the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Ozguner, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Varlık Mahallesi, Halil Sezai Erkut Caddesi Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maranto CJ, Strickland NR, Goree JH. Combined Superficial and Deep Serratus Plane Block With Bupivacaine, Dexamethasone, and Clonidine in the Treatment of a Patient With Postmastectomy Pain Syndrome: A Case Report. A A Pract. 2018 Nov 1;11(9):236-237. doi: 10.1213/XAA.0000000000000792. PMID 29794801
- [Result] Zhao J, Han F, Yang Y, Li H, Li Z. Pectoral nerve block in anesthesia for modified radical mastectomy: A meta-analysis based on randomized controlled trials. Medicine (Baltimore). 2019 May;98(18):e15423. doi: 10.1097/MD.0000000000015423. PMID 31045802
- [Result] Grape S, Jaunin E, El-Boghdadly K, Chan V, Albrecht E. Analgesic efficacy of PECS and serratus plane blocks after breast surgery: A systematic review, meta-analysis and trial sequential analysis. J Clin Anesth. 2020 Aug;63:109744. doi: 10.1016/j.jclinane.2020.109744. Epub 2020 Feb 25. PMID 32109825